CLINICAL TRIAL: NCT02107664
Title: The Palliative Radiotherapy And Inflammation Study: Palliative Radiotherapy of Bone Metastasis. Classification, Inflammatory Biomarkers, and Longitudinal Clinical Follow-up
Brief Title: The Palliative Radiotherapy And Inflammation Study - PRAIS
Acronym: PRAIS
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: European palliative care research centre (Unknown); St. Olavs Hospital (Other); Alesund Hospital (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/1126
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Neoplasm Metastasis; Bone Neoplasms
Keywords: Radiotherapy; Cachexia; Inflammation; Depression
MeSH Terms: conditions — Neoplasm Metastasis; Bone Neoplasms; Cachexia; Inflammation; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genetic and Cytokine Analyses
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Radiation therapy for bone cancer pain: The group includes all cancer diagnoses, and different fractions of RT planned.
  Interventions: Radiation: Palliative RT for bone cancer pain

INTERVENTIONS:
Radiation: Palliative RT for bone cancer pain

SUMMARY:
Radiation therapy (RT) is one of the primary treatments for bone cancer pain due to metastatic cancer disease. About 6 of 10 patients obtain pain relief from RT. There are no established predictors that can be used to select patients that respond to RT. This raises the need to identify potential clinical characteristics and biomarkers that may better select patients for RT. A similar argument can be stated for the development of cachexia; there are currently no predictors that can identify patients who will develop cachexia later in the cancer disease trajectory. Cancer symptoms can be related to inflammation. Both pain, cachexia and depression are associated with inflammation in experimental and preclinical studies . Still, the clinical data on the relationship between inflammation and pain or cachexia are sparse. This is especially true for longitudinal follow-up studies.

This study will include 1000 adult patients in a multicenter, multinational longitudinal observation study of patients who receive radiation therapy for bone cancer pain. Demographic data, clinical variables, genetic biomarkers and inflammatory substances will be assessed before start of RT. The primary analysis in the study is to identify potential predictors for pain relief from RT. During follow up the study will also explore for predictors for development of cachexia and which inflammatory substances that are associated with changes in pain intensity, depression and development of cachexia.

ELIGIBILITY:
Inclusion criteria:

* Verified cancer diagnosis (based on radiological, histological, cytological or operative evidence). Those with hematological malignancies are also eligible.
* Bone metastasis verified either by bone x-ray, bone scan, computer tomography (CT) or magnetic resonance imaging (MRI)
* Patients that are about to undergo radiotherapy with palliative intent for painful bone metastasis
* Radiotherapy should be administered within one week after baseline observations are obtained
* Age ≥18 years
* Patient is able to comply with trial procedures.

Exclusion criteria:

* Pathological fracture in long bones (e.g femora or humeral shaft fractures)
* Patients not consenting to participate in the study
* On-going RT or RT administered within the last 4 weeks
* Patients who are not able to follow the trial procedures
* Previous participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to palliative RT for bone cancer pain
Sampling Method: Non-Probability Sample
Enrollment: 580 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Pain response | 3 - 8 weeks
  Complete response implies a numeric rate scale (NRS) worst pain of zero at the treated site on an 11-point rating scale, with no concomitant increase in analgesic intake.
  Partial response is defined as either i) pain reduction of two or more at the treated site on the 11-point NRS worst pain rating scale together with no increase in analgesic intake, or ii) reduction in analgesic intake of at least 25 per cent from baseline without an increase in pain score at the treated site.
  An "intermediate response" category represents any response other than complete or partial response or pain progression

SECONDARY OUTCOMES:
Cachexia | 1 year
  Cachexia defined as a) Weight loss >5% over past 6 months (in absence of simple starvation); or b) body mass index (BMI) <20 and any degree of weight loss >2%; or c) Appendicular skeletal muscle index consistent with sarcopenia (males <7・26 kg/m2; females <5・45 kg/m2) and any degree of weight loss >2%
Depression | 1 year
  Depression symptoms last 2 weeks scored i patient Health Questionnaire (PHQ) - 9.

OTHER OUTCOMES:
Inflammatory Biomarkers | 1 year
  Change in inflammatory biomarkers during longitudinal follow-up in relation to change in pain, depression and cachexia.

CONTACTS AND LOCATIONS:
Overall Officials: Pål Klepstad, phd md, Study Director — Norwegian University of Science and Technology
Locations (3):
- Norway (3):
  - Dept of Oncology, Ålesund sjukehus, Ålesund
  - Dept of Oncology, Oslo Universitetssykehus, Oslo
  - Dept of Oncology, St Olavs Hospital, Trondheim

REFERENCES:
- [Background] Habberstad R, Froseth TCS, Aass N, Abramova T, Baas T, Morkeset ST, Caraceni A, Laird B, Boland JW, Rossi R, Garcia-Alonso E, Stensheim H, Loge JH, Hjermstad MJ, Bjerkeset E, Bye A, Lund JA, Solheim TS, Vagnildhaug OM, Brunelli C, Damas JK, Mollnes TE, Kaasa S, Klepstad P. The Palliative Radiotherapy and Inflammation Study (PRAIS) - protocol for a longitudinal observational multicenter study on patients with cancer induced bone pain. BMC Palliat Care. 2018 Sep 28;17(1):110. doi: 10.1186/s12904-018-0362-9. PMID 30266081
- [Derived] Urrizola A, Dajani O, Aass N, Bjerkeset E, Hjermstad MJ, Kaasa S, Klepstad P, Pirnat A, Raaness I, Steinsheim H, Bye A. Nutrition impact symptom monitoring and weight loss outcomes: a longitudinal radiotherapy study. BMJ Support Palliat Care. 2025 Jun 27;15(4):522-525. doi: 10.1136/spcare-2024-004939. PMID 38862183
- [Derived] Bye A, Bjerkeset E, Stensheim H, Loge JH, Hjermstad MJ, Klepstad P, Habberstad R, Kaasa S, Aass N. Benefits of Study Participation for Patients with Advanced Cancer Receiving Radiotherapy: A Prospective Observational Study. Palliat Med Rep. 2022 Nov 3;3(1):264-271. doi: 10.1089/pmr.2022.0044. eCollection 2022. PMID 36876292